CLINICAL TRIAL: NCT06414902
Title: 18F-AraG PET/CT as a Non-Invasive Imaging Biomarker for Chemoradiation Treatment Response in Esophageal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0858; NCI-2024-04295 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-FAraG PET (Experimental): Participants found to be eligible to take part in this study, participant will have a 18F-FAraG PET scan as described below. Before you start treatment, you will have standard-of-care imaging and then undergo the research 18F-FAraG PET scan. About 20 minutes before the injection of the 18F-FAraG imaging tracer, you will drink two 8-ounce bottles of water to help clear the imaging tracer from your kidneys.
  Interventions: Drug: ArabinoFuranosylGuanine [18F]F-AraG

INTERVENTIONS:
Drug: ArabinoFuranosylGuanine [18F]F-AraG — Given by IV

SUMMARY:
To learn if 18F-FAraG PET scans can find tumors in participants with esophageal cancer and predict a participant's response to treatment.

DETAILED DESCRIPTION:
Primary Objectives

* Evaluate the ability of 18F-FAraG PET imaging to detect tumors in participants with esophageal cancer;
* Evaluate 18F-FAraG PET as a predictor of pathologic complete response

Secondary Objectives

* Evaluate the correlation of 18F-FAraG PET with clinical characteristics
* Evaluate the correlation of 18F-FAraG PET with scRNA-seq data
* Evaluate tissue and blood biomarkers as predictors of treatment response and disease recurrence
* Evaluate functional imaging with 18F-FAraG PET and tissue and blood biomarkers as predictors of overall survival and disease-free survival
* Compare 18F-FAraG PET SUV update to the change in standard 18FDG-PET SUV parameters before and after chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be ≥18 years of age
2. Participants with locally advanced esophageal cancer
3. Participants with untreated documented carcinoma of the esophagus that is > 2 cm in patients who are going to receive systemic therapy concurrently with radiation as primary therapy are eligible
4. Ability to provide written informed consent in accordance with institutional policies
5. Female participants of childbearing potential must have a negative serum or urine pregnancy test within 1 week of the proposed investigational PET/CT scan(s) prior to injection of the investigational radiopharmaceutical
6. The effects of 18F-FAraG PET on the developing human fetus are unknown. For this reason and because 18F-FAraG PET agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female participants, between the onset of menses (as early as 8 years of age) and 55 years unless the participant presents with an applicable exclusionary factor which may be one of the following:

   * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
   * History of hysterectomy or bilateral salpingo-oophorectomy.
   * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
   * History of bilateral tubal ligation or another surgical sterilization procedure.
7. Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

1. Body weight ≥400 pounds or body habitus or disability that will not permit the imaging protocol to be performed
2. Pregnant or lactating females - Pregnant women are excluded from this study because 18F-FAraG PET agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with [Agent], breastfeeding should be discontinued if the mother is treated with [Agent]. These potential risks may also apply to other agents used in this study.
3. History of allergic reaction to intravenous contrast
4. eGFR<40 within 1 month prior to receiving 8F-FAraG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org